CLINICAL TRIAL: NCT02130492
Title: A Pilot Study Treatment of Malignant Tumors Using [18F] Fluorodeoxyglucose (FDG)
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Temporarily interrupted due to lack of funding: will re-open in the near future
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB# 13-382A
Record Dates: First submitted 2014-05-01; First posted 2014-05-05 (Estimated); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Advanced Cancer
Keywords: Stage IV cancers; Advanced lymphomas; Advanced sarcomas; Advanced solid tumors; Advanced cancers; Recurrent cancers; Hypermetabolic tumors
MeSH Terms: conditions — Neoplasms | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FDG arm (Experimental): Patients will receive increasing doses of FDG.
  Interventions: Radiation: FDG

INTERVENTIONS:
Radiation: FDG — The intervention arm consists of treatment with increasing doses of [18F]-Fluorodeoxyglucose.
  Other Names: [18F]-Fluorodeoxyglucose

SUMMARY:
The objectives of this Pilot study are to investigate the toxicity and safety of high doses of [18F]-Fluorodeoxyglucose (FDG) used as a therapeutic agent in patients with advanced stage IV malignant tumors that failed standard of care treatment, have a good performance status and bear radiosensitive tumors with a high [18F]-FDG uptake.

The investigators hypothesize that [18F]FDG may have a significant tumoricidal effect on cancer cells and radionuclide therapy of cancers with high doses of [18F]FDG administered as a single dose or in multiple doses (dose fractionation regimen) can be safe and well tolerated with minimal toxicities. Advantages of FDG are its uptake in many different human tumors, its short half-life (110 minutes) and the possibility to monitor its effect closely with the FDG-PET scan. The rationale for using high doses of this radiopharmaceutical agent for treatement is that most malignant lesions have accentuated glucose metabolism, which is mirrored by increased uptake of FDG. Since FDG cannot be metabolized within the cell like glucose, it is effectively confined within the cancer cells; thus, FDG treatment is potentially a novel form of targeted therapy for tumors with increased FDG uptake.

DETAILED DESCRIPTION:
Photons, electrons and protons have therapeutic use however positrons have only been used for diagnostic imaging purposes.. The energies of positrons (β+) from F-18 (0.633 MeV) and electrons (β-) from I-131 (0.606 MeV) are very close and have similar equilibrium dose constants. Since [18F]- fluorodeoxyglucose (18F-FDG) clears rapidly from circulation, administration of 37-74 BGq (1-2 Ci) of 18F-FDG is relatively safe from an internal radiation dosimetry point of view. We initiated a phase I dose escalation study to assess the safety, toxicity, and potential therapeutic utility of administering high doses of 18F-FDG delivered over a 1 to 5 day period in patients with advanced lymphomas and solid tumors refractory to standard of care treatment (SCT). There will also be a Phase 2 portion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent.
* Adults 21 years and older.
* Stage IV solid cancers and stage IV lymphomas that failed to respond to two or more regimens of standard chemotherapy.
* Life expectancy more than 3 months.
* ECOG performance status equal to or less than 2.
* Pathologically documented solid tumors and lymphoma.
* SUV in the primary tumor and/or at least one of the metastatic lesions will need to have an SUV ratio tumor to liver at least greater than 5 and the SUV in the bladder should not be above 100.
* Adequate bone marrow, hepatic and renal function as evidenced by:

  * Liver function: bilirubin < 1.5x upper limit of normal (ULN) and SGOT (AST) < 2.5x ULN.
  * Renal function: Serum creatinine <1.5 times the ULN or creatinine clearance above 50.
  * Bone marrow function: WBC above 4,000/µl; platelet count above 100,000/mm3, absolute neutrophil count above 1,500/mm3, Hemoglobin above 10 g/dl.
* Absence of brain metastases.
* No patients under the age of 21 and no pregnant or nursing women will be enrolled. Women who are not of child bearing potential, and women of child bearing potential who agree to use, while on study, an effective form of contraception and who have a negative serum pregnancy test within 72 hours prior to initial study treatment. Two forms of approved contraception measures should be used simultaneously while on trial in premenopausal women.
* Men willing to use, while on study, an effective form of contraception.
* Ability to comply with all the aspects of the protocol and to come to the follow up visits as per protocol.

Exclusion Criteria:

* Unacceptable uptakes to normal organs as determined after pre-enrollment PET imaging and serum and urinary dosimetry.
* Patients with uncontrolled diabetes.
* Patients with Stage IV lymphoma that involves the bone marrow or patients with solid tumors/ metastatic disease that involves more than 25 % of the bones.
* Patients with radioresistant tumors (i.e. melanoma).
* Patients with primary or metastatic disease to the marrow, heart or brain will be enrolled in order to prevent potential toxicity to these organs.
* Patients with neurological disorders including strokes, seizure disorder, dizziness, vertigo, preexisting grade 2 or higher neuropathy, tremors.
* Mini Mental Test score less than 24.
* Unexplained temperature > 101F or <95F for any 7 consecutive days or chronic diarrhea defined as > 3 stools/day persisting for 15 consecutive days, within the 30 days prior to treatment.
* Prior chemotherapy or surgery within one month, or prior radiotherapy within 2 months.
* Immunotherapy or biologic therapy within 1 month.
* Radiation to more than 50% of the bone marrow.
* Concurrent radiotherapy, chemotherapy. Post-menopausal women who are already using estrogens/progestins as hormone replacement therapy are permitted to enter and to continue using the hormones Tamoxifen and/or Aromatase Inhibitors will be accepted.
* Significant cardiac disease (i.e. uncontrolled high blood pressure, unstable angina, congestive heart failure, myocardial infarction within the previous year) or serious cardiac arrhythmia requiring medication.
* Active acute infection or inflammation, as determined by increased wbc and fever or abnormal CXR. Inflammation in general can cause FDG uptake that may be severe enough to be confused with malignant lesions, especially when there is granulomatous inflammation such as tuberculosis, sarcoidosis, histoplasmosis, and aspergillosis among others and patients with inflammatory disorders are excluded.
* Recent fractures within 2 months.
* Psychiatric illness/social situations that may affect the patient's compliance with the treatment.
* Current use of illicit drugs that may affect the patient's compliance with the treatment.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-05 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Serious and Non-Serious Adverse Events and Type of Serious and Non-Serious Adverse Events | Up to 1 year post administration of FDG
  Evaluate for any possible side effects related to the high doses FDG administered with therapeutic intent

SECONDARY OUTCOMES:
Efficacy Outcome Measure | Up to one year post FDG treatment
  Tumor responses in terms of size (CT scans) or FDG uptake (FDG-PET scans) will be carefully recorded and monitored using RECIST Criteria.

OTHER OUTCOMES:
FDG Dosimetry for Normal Organs, Tumors and/or Metastases | 8 hours for each patient enrolled
  Evaluate dosimetry for FDG administered at high doses

CONTACTS AND LOCATIONS:
Overall Officials: Doru Paul, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States

REFERENCES:
- [Result] Paul DM, Ghiuzeli CM, Rini J, Palestro CJ, Fung EK, Ghali M, Ben-Levi E, Prideaux A, Vallabhajosula S, Popa EC. A pilot study treatment of malignant tumors using low-dose 18F-fluorodeoxyglucose (18F-FDG). Am J Nucl Med Mol Imaging. 2020 Dec 15;10(6):334-341. eCollection 2020. PMID 33329935